CLINICAL TRIAL: NCT03462407
Title: Development and Evaluation of a Novel Imitation-based Dog Assisted Intervention, 'DIAD Training', to Increase Joint Activity and Social Wellbeing for Adolescents With Developmental Disabilities.
Brief Title: Imitation-based Dog Assisted Intervention, for Children With Developmental Disabilities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Megan MacDonald, Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7848; 1R21HD091895-01 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-03-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity; Social Responsibility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized prospectively into one of three possible groups following initial assessments and screening (e.g., eligibility), 1) 15 participants in an experimental (DAID intervention), 2) 15 control participants (dog walking), 3) 15 waitlisted control participants (true control, waitlisted for DAID one-year after post-assessment 1 of the project).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DAID (Experimental): Trained assistants will help participants train their dog to engage in imitation based dog training, using positive reinforcement training (operant conditioning) focused on physical activities.
  Interventions: Behavioral: DAID
- Dog walking (Active Comparator): Trained assistants will help children train their dog to walk on a loose leash (eliminate pulling behavior) during this period using positive training techniques. The focus of this group will be on appropriate walking behavior to facilitate enjoyable independent dog-walking at home.
  Interventions: Behavioral: Dog walking
- Control (No Intervention): This group will all own family dogs but will not participate in either intervention during year 1. All participants assigned to the waitlist will be offered the DAID intervention the subsequent summer.

INTERVENTIONS:
Behavioral: DAID — The DAID intervention group will engage in imitation based dog training, using positive reinforcement training (operant conditioning) to teach their dog to copy the physical actions they demonstrate on the command "Do it".
  Arms: DAID
Behavioral: Dog walking — Children will participate in dog walking. Trained assistants will teach the children to teach their dog basic commands. Dog walking will occur during the intervention phase and children will be encourage to walk their dogs at home.
  Arms: Dog walking

SUMMARY:
This R21 application will provide a multidisciplinary One Health approach to DAID physical activity intervention for adolescents with developmental disabilities and their family dog. The novel intervention approach includes the use of the family dog in an established dog training protocol, focused on physical activity and aimed at improving physical activity, quality of life and social wellbeing for children with and without developmental disabilities. Recent pilot work has revealed physical and social-emotional improvements in children with developmental disabilities following an animal assisted intervention. There has been relatively limited research focused on the physical activity of adolescents with developmental disabilities and there remains a critical need to develop strategies that will encourage an active lifestyle for adolescents with and without developmental disabilities. Animal assisted therapy has known positive impacts on morale and is also known to reduce depressive psychological symptoms for children and adults. Yet, traditional 'service dogs' are prohibitively expensive for many families. Dog ownership alone is known to improve health-related physical activity. Thus, a critical need exists to create physical activity interventions that are easily accessible and provide manageable home-based physical activity adherence, but that are less expensive than traditional service dogs. To achieve these goals the investigators of this project have developed the following specific aims: 1) To develop and evaluate a novel DAID dog training program to promote physical activity in children with and without developmental disabilities; 2) To determine what impact participation in a DAID dog-training program has on the child's quality of life, feelings of social wellbeing and the child-dog relationship. The long term goal of this research is to improve the lives of adolescents with and without developmental disabilities. This research supports the One Health initiative and brings together aspects of improving health related to human and animal development.

DETAILED DESCRIPTION:
Several publications have demonstrated the extent of physical activity deficits in adolescent children with DD, however very few interventions have targeted this health disparity. Not only do significant disparities exist when children with DD are compared to their peers without disabilities, but without intervention, physical activity behaviors in children with DD further decline with age. The investigators, have successfully worked together on animal assisted interventions, ultimately focused on promoting physical activity in children with disabilities. Preliminary data strongly support the conclusion that physical activity, quality of life and social wellbeing improves with a family-dog-assisted intervention. While dog-assisted interventions have become increasingly popular across applied settings, the need for further empirical evaluation is clear. Given the rapid growth of scientific knowledge in the areas of developmental disabilities, human-animal interactions and canine behavior in recent years, the development and empirical evaluation of new animal assisted intervention programs built on a solid theoretical foundation and targeted to the needs of children with DD is especially critical. In addition to the development of this intervention, we will employ an experimental design to conduct within- and between-group evaluations that will be used to assess the efficacy of the proposed DAID intervention, as well as its relative value when compared with a traditional dog walking intervention and waitlist control (true control). To further strengthen our approach, the investigators will use a combination of objective validated physical (physical activity accelerometers), self-report (Quality of Life, Dog Care Responsibility Inventory, and Pet Relationship & Friendship Scales) and behavioral measures (Child-dog/Dog-child proximity seeking, sociability and attachment) to evaluate program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Between 8- 17 years with or without a disability (per parental report)
* Has a family dog (dog in the home)

Exclusion Criteria:

* Not able to follow basic instructions/

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Physical activity Change | Baseline; Immediately post intervention (after 2- 5 weeks); one-year post intervention; a fourth immediate post-intervention for waitlisted participants who participate in the intervention (~1 year and 1 month)
  Physical activity change will be measured through accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Megan MacDonald, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will involve a small sample (45 subjects) of adolescents recruited from youth programs within Corvallis and the surrounding counties/ communities including programs targeting children with developmental disabilities. Participants must also have a family dog to participate in this study. Even with the removal of all identifiers, the investigators believe that it would be difficult to protect the identities of subjects given the small region of recruitment and disability/ age characteristics of subjects and their family dogs. Therefore, the investigators are not planning to share the data.